CLINICAL TRIAL: NCT00645593
Title: Phase II Randomized Trial of Gemcitabine and Cisplatin With or Without Cetuximab in Patients With Urothelial Carcinoma
Brief Title: Study of Gemcitabine and Cisplatin With or Without Cetuximab in Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: National Comprehensive Cancer Network (Network); Bristol-Myers Squibb (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2007.097
Record Dates: First submitted 2008-03-24; First posted 2008-03-27 (Estimated); Results first posted 2014-10-27 (Estimated); Last update posted 2016-05-23 (Estimated); Status verified 2016-04

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine; Cisplatin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1, Gemcitabine and Cisplatin (Active Comparator): Gemcitabine and Cisplatin, as described in the intervention
  Interventions: Drug: Gemcitabine,; Drug: Cisplatin
- Arm 2, Cetuximab, Gemcitabine and Cisplatin (Experimental): Gemcitabine and Cisplatin with Cetuximab, as described in the intervention
  Interventions: Drug: Gemcitabine,; Drug: Cisplatin; Drug: Cetuximab

INTERVENTIONS:
Drug: Gemcitabine, — Gemcitabine will be administered intravenously at a dose of 1000 mg/m2 on Days 1, 8 and 15 of cycle. One treatment cycle is 28 days.
  Other Names: Gemzar
Drug: Cisplatin — Cisplatin will be administered intravenously at a dose of 70 mg/m2 per institutional standards on Day 1 of each cycle.
Drug: Cetuximab — Cetuximab will be administered intravenously at a dose of 500 mg/m2 on Days 1 and 15 of each cycle. One treatment cycle is 28 days.
  Other Names: Erbitux
  Arms: Arm 2, Cetuximab, Gemcitabine and Cisplatin

SUMMARY:
This study will compare the effects, good and/or bad, of chemotherapy (Gemcitabine and Cisplatin) with or without the addition of the chemotherapy drug Cetuximab to find out which treatment is better.

DETAILED DESCRIPTION:
Urothelial cancer typically begins in the lining of the bladder, the balloon-shaped organ in the pelvic area that stores urine. Urothelial cancer can also begin in the ureter (the tube connecting the kidney and bladder), part of the kidney itself, or the urethra (the tube you pass urine out of). Some Urothelial cancers remain confined to the lining, while in other cases they spread to other areas. Treatment for these cancers varies greatly depending on the stage of disease at the time of diagnosis. Study participants in this research study will have a diagnosis of urothelial cancer that is advanced or has come back after prior therapy.

There are two standard chemotherapeutic regimens for the management of this disease. One is the combination of the drugs, methotrexate, vinblastine, doxorubicin, and cisplatin (MVAC). However the toxicities associated with this treatment regimen (side effects) is high.

The other is a combination of two drugs called Cisplatin and Gemcitabine. These drugs are also known to destroy urothelial cancer cells, and are better tolerated by patients. All study participants will receive both of these drugs.

Another anti-cancer drug called Cetuximab is known to delay or prevent tumor growth and in some cases to lead to death of cancer cells by blocking certain cellular pathways that lead to tumor development. This drug has been approved by the United States Food and Drug Administration (FDA) for the treatment of colorectal cancer and for treatment of head and neck cancers. The use of Cetuximab for the treatment of urothelial cancer is investigational in this study.

The purpose of this study is to compare the safety and efficacy of Gemcitabine and Cisplatin administered with or without the addition of Cetuximab in study participants with urothelial cancer.

This is a randomized research study. Study participants will be randomized to receive either gemcitabine and cisplatin alone or in combination with Cetuximab.

ELIGIBILITY:
Inclusion Criteria:

* Study participants will be male or female at least 18 years of age
* Study participants will have a histologic/cytologic diagnosis of urothelial carcinoma (transitional cell carcinoma; either pure or mixed histology) that is metastatic, locally recurrent, or unresectable (T4bN0 or any T, N2030)
* Study participants must have measurable disease by radiologic imaging. Study participants that have received previous radiation therapy, recovered from side effects and have not had more than 25% of the bone marrow
* Study participants must have adequate bone marrow function

Exclusion Criteria:

* Study participants may not have received previous systemic chemotherapy for the current stage of disease with the following exception: prior neoadjuvant or adjuvant chemotherapy is allowed provided it has been at least 6 months since treatment with non-cisplatin containing regimens and > 1 year since treatment with a cisplatin containing regimen
* Study participants may not have received prior therapy targeting the EGFR pathway
* Study participants may not have a history or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan
* Study participants may not have known HIV due to the intense nature of the chemotherapy in this trial
* Study subjects may not have a history of congestive heart failure (CHF), chronic renal failure, active TIAs, recent (in the last 6 months) stroke, symptomatic pulmonary embolism (PE), or myocardial infarction.
* Study participants with history of DVT or incidental or asymptomatic PE will be eligible for the study as deemed appropriate by the treating physician provided they continue prophylactic or full dose anticoagulation as per standards of care for the specific event.
* Study participants must not have a prior grade 3 or 4 severe infusion reaction to monoclonal antibodies
* Study participants may not be pregnant or breastfeeding
* Study participants may not receive concurrent treatment on another therapeutic clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2008-03; Primary Completion 2014-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maha Hussain, M.D., Principal Investigator — University of Michigan
Locations (14):
- United States (14):
  - City of Hope Cancer Center, Duarte, California
  - Kenneth J. Norris Jr. Comprehensive Cancer Center, Keck School of Medicine, University of Southern California, Los Angeles, California
  - Stanford University, Stanford, California
  - Robert H. Lurie Comprehensive Cancer Center, Center of Northwestern University, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Hussain M, Daignault S, Agarwal N, Grivas PD, Siefker-Radtke AO, Puzanov I, MacVicar GR, Levine EG, Srinivas S, Twardowski P, Eisenberger MA, Quinn DI, Vaishampayan UN, Yu EY, Dawsey S, Day KC, Day ML, Al-Hawary M, Smith DC. A randomized phase 2 trial of gemcitabine/cisplatin with or without cetuximab in patients with advanced urothelial carcinoma. Cancer. 2014 Sep 1;120(17):2684-93. doi: 10.1002/cncr.28767. Epub 2014 May 6. PMID 24802654

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1, Gemcitabine and Cisplatin: Gemcitabine, Cisplatin: Cisplatin will be administered intravenously at a dose of 70 mg/m2 per institutional standards on Day 1 of each cycle. Gemcitabine will be administered intravenously at a dose of 1000 mg/m2 on Days 1, 8 and 15 of cycle. One treatment cycle is 28 days.
- Arm 2, Cetuximab, Gemcitabine and Cisplatin: Gemcitabine, Cisplatin and Cetuximab: Cisplatin will be administered intravenously at a dose of 70 mg/m2 per institutional standards on Day 1 of each cycle. Gemcitabine will be administered intravenously at a dose of 800 mg/m2 on Days 1, 8 and 15 of cycle. Cetuximab will be administered intravenously at a dose of 500 mg/m2 on Days 1 and 15 of each cycle. One treatment cycle is 28 days.
Period: Overall Study
Arm/Group | Arm 1, Gemcitabine and Cisplatin | Arm 2, Cetuximab, Gemcitabine and Cisplatin
Started | 29 | 60
Completed | 28 | 60
Not Completed | 1 | 0
Not completed — Later found to be ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: Although 89 patients were enrolled, only 88 patients were analyzed. 1 patient was randomized to arm A, was treated, and developed grade 4 neutropenia but was found to be ineligible upon histology review and was removed from the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1, Gemcitabine and Cisplatin | Arm 2, Cetuximab, Gemcitabine and Cisplatin | Total
Number analyzed (Participants) | 28 | 60 | 88
Age, Continuous [Median (Full Range); unit: years] | 65.8 [41 to 79.9] | 60.9 [32.8 to 79.4] | 61 [32 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 14 | 19
  Male | 23 | 46 | 69
ECOG performance status [Number; unit: participants] — The Eastern Cooperative Oncology Group (ECOG) performance status is an attempt to quantify cancer patients' general well-being and activities of daily life. The scoring system runs from 0 to 5 where 0 represents perfect health and 5 represents death.
  participants
    0 | 18 | 33 | 51
    1 | 8 | 26 | 34
    2 | 2 | 1 | 3
Bladder primary [Number; unit: participants] — Number of participants with cancer that originated within the bladder.
  participants | 20 | 45 | 65
Distant metastasis [Number; unit: participants] — The number of participants presenting with distant metastasis.
  participants | 26 | 54 | 80
Local recurrence [Number; unit: participants] — The number of participants presenting with local recurrence.
  participants | 1 | 2 | 3
Unresectable disease [Number; unit: participants] — The number of participants presenting with unresectable disease.
  participants | 1 | 4 | 5
Prior cystectomy or nephroureterectomy [Number; unit: participants] — The number of participants that have had a prior cystectomy or nephroureterectomy.
  participants | 10 | 13 | 23
Primary in place [Number; unit: participants] — The area of primary cancer (where the cancer originated) remains intact and has not been excised.
  participants | 18 | 47 | 65
Prior neoadjuvant or or adjuvant chemotherapy [Number; unit: participants] | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants That Respond to Treatment in Arm 1 and Arm 2
Description: The primary objective is to compare the overall response rate of participants with locally advanced or metastatic urothelial carcinoma treated with gemcitabine and cisplatin with or without cetuximab.
  Overall response rate is defined as the percentage of participants that experience Complete Response (CR) (Disappearance of all target lesions) or Partial Response (PR) (>=30% decrease in the sum of the longest diameter of target lesions).
Time Frame: 3 years
Population: 29 patients were enrolled and randomized to arm 1 and 60 patients were enrolled and randomized to arm 2. 1 patient from arm 1 was found to be ineligible and 3 patients from arm 2 withdrew consent (1 prior to treatment and 2 prior to 4 weeks of treatment). Only 28 patients from arm 1 and 57 patients from arm 2 were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1, Gemcitabine and Cisplatin | Arm 2, Cetuximab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 28 | 57
percentage of participants | 57.1 [37 to 76] | 61.4 [48 to 74]

2. Secondary Outcome: The Number of Grade 3 to 5 Adverse Events Experienced by Arm 1 and Arm 2
Description: One of the secondary outcomes was to assess the safety and tolerability of treatment for both arms.
  The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 were utilized for adverse event reporting.
Time Frame: 3 years
Population: Although 60 participants were enrolled and randomized to arm 2, 1 participant withdrew consent prior to treatment and was therefore excluded from toxicity analysis.
Measure: Number; unit: adverse events
Arm/Group | Arm 1, Gemcitabine and Cisplatin | Arm 2, Cetuximab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 28 | 59
adverse events | 75 | 83

3. Secondary Outcome: Median Progression-free Survival Time in Months
Description: Progressive disease is defined as at least a 20% increase in the sum of the longest diameter of target lesions.
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1, Gemcitabine and Cisplatin | Arm 2, Cetuximab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 28 | 57
months | 8.5 [5.7 to 10.4] | 7.6 [6.1 to 8.7]

4. Secondary Outcome: Median Overall Survival in Months
Description: Median overall survival in months is provided. One participant who progressed from chemotherapy in arm 1 received cyclophosphamide and achieved long-term disease control therefore there is no upper limit for the 95% confidence interval.
Time Frame: 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm 1, Gemcitabine and Cisplatin | Arm 2, Cetuximab, Gemcitabine and Cisplatin
Number analyzed (Participants) | 28 | 57
Months | 17.4 [12.8 to NA] — One participant who progressed from chemotherapy in arm 1 received cyclophosphamide and achieved long-term disease control therefore there is no upper limit for the 95% confidence interval. | 14.3 [11.6 to 22.2]

ADVERSE EVENTS:
Arm/Group | Arm 1, Gemcitabine and Cisplatin | Arm 2, Cetuximab, Gemcitabine and Cisplatin
Serious Adverse Events (participants affected / at risk) | 16/29 | 36/60
Other Adverse Events (participants affected / at risk) | 29/29 | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Gemcitabine and Cisplatin (N=29) | Arm 2, Cetuximab, Gemcitabine and Cisplatin (N=60)
CNS cerebrovascular ischemia (Vascular disorders) | 1 (1) | 2 (2)
Confusion (Nervous system disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Febrile neutropenia (fever of unknown origin without documented infection) (General disorders) | 2 (2) | 2 (2)
Hemorrhage, GI (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 2 (2) | 1 (1)
Infection - Other (Infections and infestations) | 1 (1) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 3 (3) | 7 (7)
Leukocytes (total WBC) (Investigations) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (7)
Neurology - Other (Nervous system disorders) | 1 (1) | 0 (0)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 5 (5) | 8 (10)
Pain (General disorders) | 2 (2) | 5 (5)
Platelets (Investigations) | 1 (3) | 7 (11)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 3 (3) | 7 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 1 (1)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 1 (1)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ataxia (incoordination) (Nervous system disorders) | 0 (0) | 2 (2)
Cardiac General - Other (Cardiac disorders) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion (Nervous system disorders) | 0 (0) | 1 (3)
Death not associated with CTCAE term (General disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Edema: limb (General disorders) | 0 (0) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 (0) | 3 (4)
Fever (in the absence of neutropenia) (General disorders) | 0 (0) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Hemorrhage, GU (Renal and urinary disorders) | 0 (0) | 1 (1)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 3 (3)
Insomnia (Nervous system disorders) | 0 (0) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 3 (5)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neuropathy: motor (Nervous system disorders) | 0 (0) | 2 (2)
Neuropathy: sensory (Nervous system disorders) | 0 (0) | 1 (1)
Obstruction, GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstruction, GU (Renal and urinary disorders) | 0 (0) | 1 (1)
Peripheral arterial ischemia (Vascular disorders) | 0 (0) | 1 (1)
Pulmonary/Upper Respiratory - Other (Specify) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Syncope (fainting) (Nervous system disorders) | 0 (0) | 1 (1)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 6 (7)
Typhlitis (cecal inflammation) (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulcer, GI (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1, Gemcitabine and Cisplatin (N=29) | Arm 2, Cetuximab, Gemcitabine and Cisplatin (N=60)
Albumin, serum-low (hypoalbuminemia) (Investigations) | 8 (12) | 13 (41)
Anorexia (Metabolism and nutrition disorders) | 15 (18) | 27 (44)
Constipation (Gastrointestinal disorders) | 14 (23) | 22 (35)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (19)
Creatinine (Investigations) | 10 (39) | 16 (40)
Dehydration (Metabolism and nutrition disorders) | 8 (10) | 15 (19)
Diarrhea (Gastrointestinal disorders) | 9 (15) | 20 (42)
Dizziness (Nervous system disorders) | 5 (6) | 16 (32)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 12 (16)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 23 (67) | 51 (146)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 13 (43) | 20 (96)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5 (5) | 13 (13)
Anemia (Blood and lymphatic system disorders) | 22 (54) | 37 (139)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 11 (13) | 28 (31)
Leukocytes (total WBC) (Investigations) | 12 (30) | 31 (114)
Lymphopenia (Investigations) | 6 (17) | 19 (100)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6 (18) | 31 (132)
Mood alteration (Nervous system disorders) | 7 (9) | 13 (20)
Nausea (Gastrointestinal disorders) | 17 (43) | 38 (71)
Neuropathy: sensory (Nervous system disorders) | 8 (10) | 16 (22)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 18 (44) | 36 (100)
Pain (General disorders) | 29 (46) | 60 (136)
Pain - Other (General disorders) | 6 (7) | 8 (12)
Platelets (Investigations) | 26 (96) | 45 (162)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 7 (15) | 11 (32)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 7 (23) | 7 (11)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 9 (11) | 14 (19)
Tinnitus (Ear and labyrinth disorders) | 5 (6) | 0 (0)
Urinary frequency/urgency (Renal and urinary disorders) | 5 (8) | 0 (0)
Vomiting (Gastrointestinal disorders) | 8 (14) | 20 (29)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 0 (0) | 12 (36)
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 0 (0) | 11 (38)
Alkaline phosphatase (Investigations) | 0 (0) | 8 (22)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 0 (0) | 5 (5)
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 0 (0) | 6 (9)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 (0) | 11 (18)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 15 (19)
Dermatology/Skin - Other (Specify) (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (20)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 16 (22)
Edema: limb (General disorders) | 0 (0) | 16 (22)
Fever (in the absence of neutropenia) (General disorders) | 0 (0) | 12 (18)
Heartburn/dyspepsia (Gastrointestinal disorders) | 0 (0) | 15 (22)
Hemorrhage, GU (Renal and urinary disorders) | 0 (0) | 8 (8)
Hemorrhage, pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (7)
Hypertension (Cardiac disorders) | 0 (0) | 6 (9)
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils (Infections and infestations) | 0 (0) | 8 (8)
Infection - Other (Infections and infestations) | 0 (0) | 6 (8)
Infection with unknown ANC (Infections and infestations) | 0 (0) | 10 (11)
Insomnia (Nervous system disorders) | 0 (0) | 6 (6)
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 0 (0) | 6 (18)
Mucositis/stomatitis (clinical exam) (Gastrointestinal disorders) | 0 (0) | 9 (11)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 0 (0) | 7 (7)
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (9)
Nail changes (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (9)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 (0) | 11 (23)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 27 (85)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 33 (118)
Rigors/chills (General disorders) | 0 (0) | 9 (12)
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 0 (0) | 5 (9)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 (0) | 21 (49)
Supraventricular and nodal arrhythmia (Cardiac disorders) | 0 (0) | 9 (11)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 0 (0) | 8 (9)
Thrombosis/thrombus/embolism (Vascular disorders) | 0 (0) | 9 (10)
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (6)
Weight loss (Investigations) | 0 (0) | 11 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes